CLINICAL TRIAL: NCT07029828
Title: A LONG-TERM, DOUBLE-BLIND EXTENSION STUDY TO INVESTIGATE THE SAFETY AND EFFICACY OF RITLECITINIB IN PARTICIPANTS WITH SEVERE ALOPECIA AREATA WHO PREVIOUSLY COMPLETED STUDIES B7981027 OR B7981031
Brief Title: A Long-Term Study to Learn About The Study Medicine Called Ritlecitinib in Children With Severe Alopecia Areata.
Acronym: B7981028
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981028; 2024-515439-31-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Severe Alopecia Areata
Keywords: Alopecia Areata; Children; Ritlecitinib; Long-term extension study
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ritlecitinib higher dose (Experimental): Participants will receive 1 ritlecitinib higher dose capsule once a day (QD) and 1 placebo lower dose capsule QD orally for up to 3 years.
  Participants who meet the protocol-defined treatment discontinuation criteria based on not achieving the required efficacy threshold will be switched to placebo but will remain in the study.
  Those participants will receive 1 placebo higher dose capsule QD and 1 placebo lower dose capsule QD.
  Interventions: Drug: Ritlecitinib higher dose
- Ritlecitinib lower dose (Experimental): Participants will receive 1 ritlecitinib lower dose capsule once a day (QD) and 1 placebo higher dose capsule QD orally for up to 3 years.
  Participants who meet the protocol-defined treatment discontinuation criteria based on not achieving the required efficacy threshold will be switched to placebo but will remain in the study.
  Those participants will receive 1 placebo higher dose capsule QD and 1 placebo lower dose capsule QD.
  Interventions: Drug: Ritlecitinib lower dose

INTERVENTIONS:
Drug: Ritlecitinib higher dose — Study intervention will be provided as oral capsules centrally by the sponsor in HDPE bottles.
  Arms: Ritlecitinib higher dose
Drug: Ritlecitinib lower dose — Study intervention will be provided as oral capsules centrally by the sponsor in HDPE bottles.
  Arms: Ritlecitinib lower dose

SUMMARY:
The purpose of this clinical trial is to learn about long-term safety and long-term effects of the study medicine (called ritlecitinib) for the potential treatment of severe alopecia areata, a condition that causes hair loss.

This study is seeking participants who have:

* previously completed one of Pfizer's pediatric studies for Alopecia Areata (B7981027 or B7981031).
* at least 50% scalp hair loss due to alopecia areata (for participants enrolling from the study B7981031).
* received varicella vaccination (2 doses) or have been infected by varicella zoster virus before based on blood test reports.

All participants in this study will receive the study medicine (ritlecitinib). Participants who received ritlecitinib higher or lower doses in the parent Study B7981027 will continue receiving the same ritlecitinib dose in this trial.

Participants who received placebo in the parent Study B7981027 and all participants from parent Study B7981031 will receive either higher or lower dose of ritlecitinib in this trial.

The study medicine is a capsule that is taken by mouth. It is taken 1 time each day at home.

The study will help see if ritlecitinib is safe and effective. Participants will take part in this study for a duration of up to 3 years (36 months). During this time, they will have 17 study visits at the study clinic. The study team will also call participants once a month over the phone.

DETAILED DESCRIPTION:
Study B7981028 is a Phase 3 long-term, double-blind extension study to evaluate the safety and efficacy of ritlecitinib in participants with severe alopecia areata (AA) who have completed previous ritlecitinib studies B7981031 or B7981027 and are eligible to enroll for B7981028 study.

The primary objective of this study is to evaluate the long-term safety and tolerability of ritlecitinib in pediatric participants with severe AA who have completed the studies B7981027 or B7981031. The secondary objectives of this study are to evaluate the long-term efficacy of ritlecitinib, durability of response and effect of ritlecitinib on patient centered outcomes.

All participants in this study will receive ritlecitinib higher or lower dose for up to an additional 3 years following completion of either of the prior parent studies. Participants who received higher or lower doses in the parent Study B7981027 will continue receiving the same ritlecitinib dose in Study B7981028. Participants who received placebo in the parent Study B7981027 and all participants from parent Study B7981031 will be randomized at a 1:1 ratio to receive higher or lower dose of ritlecitinib in Study B7981028.

At least 140 participants evaluable for primary analysis will be enrolled in Study B7981028.

Participants will be evaluated for treatment continuation criteria at Months 3 and 6 (for those who were previously assigned to active treatment in parent Study B7981027) and at Months 9 and 12 in Study B7981028 (for those who previously completed Study B7981031 or were assigned to placebo in the parent Study B7981027). Ritlecitinib treatment will be discontinued for any participant who does not meet the study treatment continuation criteria.

Safety monitoring will be performed to identify and monitor the known and potential risks of ritlecitinib.

The efficacy assessments include Severity of Alopecia Tool (SALT), eyebrow and eyelash assessments. Patient reported outcomes including Patient's Global Impression of Change (PGI-C), Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy - Anxiety Short Form 8a and Depressive Symptoms Short Form 6a, Behavior Rating Inventory of Executive Function®, Second Edition (BRIEF®2), and modified Children's Dermatology Life Quality Index (CDLQI) will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with alopecia areata (AA) (including alopecia totalis [AT] and alopecia universalis [AU]) who completed the studies B7981027 or B7981031.
2. For participants originating from Study B7981031: At least 50% scalp hair loss due to AA (ie, a SALT score of ≥50) at both the Screening and Baseline visits.

Exclusion Criteria:

1. Exclusion criteria for participants originating from Study B7981027 with ≤ 30 Days between last dose in Study B7981027 and first visit of Study B7981028

   1. During Study B7981027 or in the period between the last dose of study intervention in Study B7981027 and the first dose of study intervention of Study B7981028, presence of safety events that would require permanent discontinuation based on the B7981028 protocol.
   2. Study participants discontinued from Study B7981027 due to issues other than safety-related events and considered by the investigator for enrolment in Study B7981028 must have resolution of the issue(s) resulting in discontinuation from the parent study prior to enrolment in Study B7981028.
2. Exclusion criteria for participants originating from Study B7981031 or from Study B7981027 with >30 Days between last dose in Study B7981027 and first visit of Study B7981028

   1. During Study B7981031 or Study B7981027 or in the period between the last dose of study intervention in Study B7981031 or Study B7981027 and the first dose of study intervention of Study B7981028, presence of safety events that would require permanent discontinuation based on the B7981028 protocol.
   2. Any present malignancies or history of malignancies or lymphoproliferative disorders.
   3. Evidence of untreated or inadequately treated active or latent Mycobacterium tuberculosis (TB) infection, history (one or more episodes) of severe or serious cytomegalovirus (CMV), herpes zoster (shingles) or disseminated herpes simplex, infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).

      -

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2030-06-26 (Estimated); Study Completion 2030-06-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs). | From the time participant signs informed consent/assent, through and including a minimum of 28 calendar days after the last administration of the study intervention (up to approximately 3 years).
Incidence of Serious Adverse Events (SAEs) and AEs leading to permanent discontinuation from the study. | From the time participant signs informed consent/assent, through and including a minimum of 28 calendar days after the last administration of the study intervention (up to approximately 3 years).

SECONDARY OUTCOMES:
Proportion of participants achieving absolute Severity of Alopecia Tool (SALT) score ≤10. | Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
Proportion of participants achieving absolute SALT score ≤20. | Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
Change from baseline (CFB) in SALT score. | Baseline, Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
Proportion of participants achieving at least 2 grade improvement or a score of 3 in eyebrow assessment (EBA) score in participants with an abnormal EBA at baseline. | Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
Proportion of participants achieving at least 2 grade improvement or a score of 3 in eyelash assessment (ELA) score in participants with an abnormal ELA at baseline. | Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
Proportion of participants achieving Patient Global Impression of Change (PGI-C) response defined as a score of "moderately improved" or "greatly improved". | Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
CFB in PROMIS Parent Proxy Anxiety Symptoms T-score. | Baseline, Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
CFB in Behavior Rating Inventory of Executive Function (BRIEF®2) T-scores for the 3 index scores (Behavior Regulation Index (BRI), Emotion Regulation Index (ERI), Cognitive Regulation Index (CRI)). | Baseline, Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
CFB in modified Children's Dermatology Life Quality Index (CDLQI) total score. | Baseline, Months 3,6,9,12,15,18,21,24,27,30,33 and 36.
CFB in Wechsler Intelligence Scale for Children® Fifth Edition (WISC-V). | Baseline, Month 36

OTHER OUTCOMES:
CFB in Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Depressive Symptoms T-score. | Baseline, Months 3,6,9,12,15,18,21,24,27,30,33 and 36.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pediatric Skin Research, Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Northwest Dermatology Institute, Portland, Oregon
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981028